CLINICAL TRIAL: NCT01424683
Title: Development of a Method for Converting VAS Scores for Pain and Mobility to EQ-5D Answers
Brief Title: Development of a Method for Converting Visual Analogue Scale (VAS) Scores for Pain and Mobility to EQ-5D Answers
Status: Completed | Type: Observational
Sponsor: Lars Oddershede (Other)
Responsible Party: Sponsor-Investigator, Lars Oddershede, MMSc (master of medical science), Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Other Study IDs: Oddershede-1
Record Dates: First submitted 2011-08-25; First posted 2011-08-29 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Cardiovascular Diseases
Keywords: Qol; Quality of life; VAS; Visual Analogue Scale; CABG; Coronary Artery Bypass Graft; Qol conversion; post hoc HTA
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Endoscopic Vein Harvest (EVH): A short saphenous vein segment is commonly used as a conduit for coronary artery bypass grafting (CABG), and clinicians must decide whether to obtain it by performing a traditional open vein harvest (OVH) or by performing an endoscopic vein harvest (EVH).
- Open Vein Harvest (OVH): A short saphenous vein segment is commonly used as a conduit for coronary artery bypass grafting (CABG), and clinicians must decide whether to obtain it by performing a traditional open vein harvest (OVH) or by performing an endoscopic vein harvest (EVH).

SUMMARY:
The objective of this study is to investigate how mobility and pain scores, measured on a Visual Analogue Scale (VAS), correspond to patients' EuroQol-5Dimensions-3Levels (EQ-5D-3L) answers on pain and mobility. In addition, the investigators want to evaluate patients' undergoing Coronary Artery Bypass Grafting (CABG) quality of life postoperatively, depending on the vein harvesting method used.

DETAILED DESCRIPTION:
Many health economic researchers prefer that a treatments effect is measured in the quantity and quality of life (Qol) the treatment provides. This enables them to calculate effect in the generic Quality Adjusted Life-Years (QALYs). Patients' Qol can be estimates by having patients' answer the EQ-5D-3L questionnaire. However, when performing a post hoc health economic evaluation, data is often incomplete. Often there is no information available regarding the patients' Qol and some health economic researchers therefore resort to various conversions of other measurements of effect to Qol. Such conversions thereby enable them to calculate effect in QALYs even though they had incomplete information. However, no method has been developed for converting eg. VAS pain scores to Qol and the methods currently used are arbitrary. With this study the investigators wish to develop such a method and in the process evaluate our own arbitrary Qol conversion from a prior study by asking the same type of patients. The study is an observational study with no intervention.

ELIGIBILITY:
Inclusion Criteria:

* Elective CABG patients
* Use of a vein segment for conduit during CABG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing CABG
Sampling Method: Non-Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2011-08; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
The distribution of answers to EQ-5D-3L sub-questions on a 100mm VAS for each sub-question. | Approximately five days postoperatively
  The investigators wish to investigate how patients scoring "no pain or discomfort", "moderate pain or discomfort" and "extreme pain or discomfort" on the EQ-5D questionnaire score their pain on a 100mm VAS of pain. The same is done for the four other sub-questions in the EQ-5D, eg. how do patients score their mobility on a 100mm VAS of mobility if they score "no problems in walking about", "some problems in walking about" or "confined to bed" on the EQ-5D. (see citations for similar study setups)

SECONDARY OUTCOMES:
Quality of life (Qol) | approximately 30 days
  The investigators will obtain 3 measurements from each patient and are therefore able to evaluate the change in Qol from baseline to approximately 30 days postoperatively in a group of elective bypass patients. Investigators hereby aim to find the incremental Qol. The patient group will be segmented on whether they underwent endoscopic or open vein harvest during their surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Jan J Andreasen, MD, PhD, Study Director — Department of Cardiothoracic Surgery, Center for Cardiovascular Research, Aalborg Hospital, Aarhus University Hospital; Lars Oddershede, MMSc, Principal Investigator — Department of Cardiothoracic Surgery, Center for Cardiovascular Research, Aalborg Hospital, Aarhus University Hospital
Locations (1):
- Aalborg Hospital, Aalborg, Region Nord, Denmark

REFERENCES:
- [Background] Jensen MP, Chen C, Brugger AM. Interpretation of visual analog scale ratings and change scores: a reanalysis of two clinical trials of postoperative pain. J Pain. 2003 Sep;4(7):407-14. doi: 10.1016/s1526-5900(03)00716-8. PMID 14622683
- [Background] Collins SL, Moore RA, McQuay HJ. The visual analogue pain intensity scale: what is moderate pain in millimetres? Pain. 1997 Aug;72(1-2):95-7. doi: 10.1016/s0304-3959(97)00005-5. PMID 9272792